CLINICAL TRIAL: NCT07009535
Title: Associations Apnoea Hypopnoea Index (AHI) and Malocclusions in Growing Patients With Maxillary Constriction: a Prospective Clinical Study.
Brief Title: Associations Apnoea Hypopnoea Index (AHI) and Malocclusions in Growing Patients With Maxillary Constriction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-AHIO2AIRWAYS
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Apnea, Obstructive Sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients between 6 and 12 years with maxillary constriction (intermolar distance < 31 mm) requiring rapid palatal expander therapy and with AHI > 1
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Assessment of AHI index and pO2 in pediatric patients

SUMMARY:
The aim of this prospective clinical study is to evaluate the association between the Apnoea Hypopnoea Index (AHI) and the type of malocclusion in pediatric patients with maxillary constriction. Malocclusion will be assessed through clinical examination and cephalometric analysis, which will also include an evaluation of the airway. Additionally, the study aims to assess potential changes in OSAS symptoms in patients undergoing orthopedic-orthodontic treatment with maxillary expansion. The AHI assessment will be conducted using nocturnal cardiorespiratory monitoring.

DETAILED DESCRIPTION:
This observational study aims to evaluate possible associations between data obtained from cardiorespiratory monitoring, clinical examination, and cephalometric analysis in patients with maxillary constriction. First, patients aged 6 to 12 years who present to the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic, and Pediatric Sciences of the University of Pavia will undergo a clinical examination to assess the presence of malocclusions. If malocclusions are identified, the necessary records for the patient's diagnostic-therapeutic assessment will be collected. During the initial visit, parents will also be asked to complete the PSQ-SRBD questionnaire (1) (Appendix A), which serves as a screening test for OSAS. Subsequently, the transpalatal width will be measured on plaster or digital models by evaluating the intermolar distance. According to McNamara, this value in mixed dentition without crowding or spacing ranges between 34 and 36 mm (2), while it is less than 31 mm in cases of crowding, indicating the need for orthopedic or surgical expansion (3). In this study, a cut-off value of 31 mm was used to select the sample with maxillary constriction. If such a malocclusion is present, the operators will verify whether the patient meets the study's inclusion criteria. Cephalometric analysis will be performed on lateral cranial radiographs, focusing on craniofacial characteristics and upper airway measurements, as detailed later in the protocol. The selected children will then be referred to the Sleep Medicine Center at the Mondino Foundation for cardiorespiratory monitoring (AHI). Data from the polygraphic examination, cephalometric analysis, and clinical evaluation will be compared using statistical analysis. If the patient is diagnosed with OSAS (AHI >1) and requires palatal expansion, cardiorespiratory monitoring, clinical evaluation, and cephalometric analysis will be repeated after treatment with an expander and compared with the initial data.

ELIGIBILITY:
Inclusion Criteria:

* mixed dentition
* transversal skeletal constriction of the upper jaw, with or without cross-bite
* Tonsillar grade I-III according to Mallampati classification

Exclusion Criteria:

* Previous orthodontic treatment
* Previous adenoidectomy, tonsillectomy, or any surgical interventions of the upper airways;
* Tonsillar grade IV
* Presence of remote or familial pathologies;
* Presence of syndromes or forms of disability

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  The number of apneas and/or hypopneas per hour of recording. It is considered mild OSAS if AHI is between 1 and 5; moderate OSAS if AHI is between 5 and 10; severe OSAS if AHI is greater than 10.

SECONDARY OUTCOMES:
SNA Angle | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Determined by the intersection of the sellar plane (SN) with the N-point A line; it indicates the anteroposterior position of the maxilla relative to the cranial base. Mean value: 82° ± 2°.
SNB Angle | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Determined by the intersection of the sellar plane (SN) with the N-point B line; it indicates the anteroposterior position of the mandible relative to the cranial base. Mean value: 80° ± 2°.
ANB Angle | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Determined by the intersection of the N-point A line with the N-point B line; it indicates the anteroposterior relationship between the maxilla and mandible. The discrepancy identified by this angle defines the skeletal class. Mean value: 2° ± 2°.
Cranio-mandibular Angle (SN^GoGn) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Determined by the intersection of the sellar plane (SN) with the mandibular plane (GoGn); it indicates the type of vertical facial growth of the subject. Mean value: 32° ± 5°.
Intermaxillary Angle (ANS-PNS^GoGn) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Determined by the intersection of the bipupillary plane (ANS-PNS) with the mandibular plane (GoGn); it indicates the degree of divergence of the mandible relative to the cranial base. Mean value: 20° ± 5°.
Ad1-SNP | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Linear distance between SNP and the closest point on the posterior wall of the pharynx along the line connecting SNP-Ba.
Ad2-SNP | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Linear distance between SNP and the closest point on the posterior wall of the pharynx measured through the perpendicular line to the connecting S-Ba from the SNP point.
MPP-SPAS | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Superior pharyngeal space. Connects the point MPP (midpoint of the pharyngeal side of the velum placed on a line perpendicular to the line connecting SNP-U1) and the point SPAS (point on the posterior wall of the pharynx determined by a perpendicular line to the posterior pharyngeal wall passing through MPP).
U1-U2 | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Middle pharyngeal space: connects U1 (tip of the soft palate) and U2 (point on the posterior wall of the pharynx determined by a perpendicular line to the posterior pharyngeal wall passing through U1).
T1-T2 | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Inferior pharyngeal space: distance between point T1 (intersection between the tongue base and the lower margin of the mandible) and point T2 (projection of point T1 on the posterior wall of the pharynx along the parallel to the line Go-Ba).
Thickness (MPP-MPA) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Connects the points MPP (midpoint of the pharyngeal side of the velum, placed on a line perpendicular to the line connecting SNP with U1) and MPA (point on the oral side of the velum placed on a line perpendicular to the line connecting SNP with U1).
Length (U-SNP) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Distance between the tip of the soft palate (U1) and the posterior nasal spine (SNP).
MPH | Baseline (T0) and after 1 year of treatment with RPE (T1)
  Distance between point H1 (most cranial point of the hyoid bone) and point H2 (projection of point H1 on the perpendicular to the lower margin of the mandible - GoGn).
Molar Class | Baseline (T0) and after 1 year of treatment with RPE (T1)
  * Class I molar: The mesiobuccal cusp of the upper first molar contacts the vestibular groove of the lower first molar.
  * Class II molar: The mesiobuccal cusp of the upper first molar occludes mesially to the vestibular groove of the lower first molar.
  * Class III molar: The mesiobuccal cusp of the upper first molar occludes distally to the vestibular groove of the lower first molar.
Overjet | Baseline (T0) and after 1 year of treatment with RPE (T1)
  The distance, in the sagittal plane, between the upper and lower incisal edges. Mean value: 2 ± 2 mm. If > 2 mm, it is considered "increased"; if < 2 mm, it is considered "reduced".
Overbite | Baseline (T0) and after 1 year of treatment with RPE (T1)
  The distance, in the vertical plane, between the upper and lower incisal edges. Mean value: 2 ± 2 mm. If > 2 mm, it is considered "increased"; if < 2 mm, it is considered "reduced".
Oxygen Saturation (Nadir SpO2) | Baseline (T0) and after 1 year of treatment with RPE (T1)
  The minimum percentage of oxygen-saturated hemoglobin at the time of measurement. SpO2 values are as follows: between 86% and 91% in mild OSAS, between 76% and 85% in moderate OSAS, and less than 75% in severe OSAS.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — Associate Professor
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.